CLINICAL TRIAL: NCT02748993
Title: A Randomized, Double-blind, Placebo-Controlled, Parallel Study to Investigate the Safety, Tolerability, Systemic Exposure and Efficacy of PAC-14028 in Children With Mild to Moderate Pediatric Atopic Dermatitis
Brief Title: A Study to Evaluate the Safety and Efficacy of PAC-14028 Cream in Pediatric Atopic Dermatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amorepacific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP-TRPV1_PII-05
Record Dates: First submitted 2016-04-20; First posted 2016-04-22 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PAC-14028 Cream 0.1% (Experimental): PAC-14028 Cream 0.1%, Twice daily for 4 weeks
  Interventions: Drug: PAC-14028 Cream 0.1%
- PAC-14028 Cream 0.3% (Experimental): PAC-14028 Cream 0.3%, Twice daily for 4 weeks
  Interventions: Drug: PAC-14028 Cream 0.3%
- PAC-14028 Cream 1.0% (Experimental): PAC-14028 Cream 1.0%, Twice daily for 4 weeks
  Interventions: Drug: PAC-14028 Cream 1.0%
- PAC-14028 Cream Vehicle (Placebo Comparator): PAC-14028 Cream Vehicle, twice daily for 4 weeks
  Interventions: Drug: PAC-14028 Cream Vehicle

INTERVENTIONS:
Drug: PAC-14028 Cream 0.1% — Topical application
  Arms: PAC-14028 Cream 0.1%
Drug: PAC-14028 Cream 0.3% — Topical application
  Arms: PAC-14028 Cream 0.3%
Drug: PAC-14028 Cream 1.0% — Topical application
  Arms: PAC-14028 Cream 1.0%
Drug: PAC-14028 Cream Vehicle — Topical application
  Arms: PAC-14028 Cream Vehicle

SUMMARY:
This is a phase 1 and 2 study to assess the safety and efficacy of PAC-14028 cream in children with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 24 months - 12 years
* Who was diagnosed with Atopic Dermatitis according to Haniffin and Rajka criteria, whose affected BSA is over 5% and IGA score is 2 (mild) to 3 (moderate).
* Who has applied stable amount of emollients daily before baseline visit
* Who voluntarily agreed to participate in the study and signed an informed consent form.

Exclusion Criteria:

* Who has skin diseases other than atopic dermatitis or scar in the affected area which can affect the study, determined by the study investigators.
* Who has clinically significant medical history or diseases involving liver, kidney, neurological system, psychial disorder that can affect study results.
* Who has used systemic steroids, antibiotics, immunosuppressants, or received photochemical therapy within 28 days before study drug administration.
* Who has used topical steroids, immunosuppressants or antibiotics to treat atopic dermatitis within 14 days before study drug administration.
* Who has used or is expected to inevitably use prohibited concomitant medications during the study.
* Women who is pregnant /breast-feeding, or who has childbearing potential and does not use available contraceptives.
* Who has dosed other study medications within 30 days before screening.
* Who is determined ineligible for study participation by investigators for any other reasons.

Ages: 24 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2016-03; Primary Completion 2018-09 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Success rate of Investigator's Global Assessment (IGA) | 4 weeks
  % of patients with IGA score of 0 (clear) or 1 (almost clear)
Blood concentrations of PAC-14028 | Day 1, Day 28
  Blood concentrations of PAC-14028

SECONDARY OUTCOMES:
Change of IGA (Investigator's Global Assessment) | 1, 2, 4 week(s)
  Change of IGA score from baseline
Change of SCORAD (Severity Scoring of Atopic Dermatitis) | 1, 2, 4 week(s)
  Change of SCORAD from baseline
% Change of EASI (Eczema Area and Severity Index) | 1, 2, 4 week(s)
Patient satisfaction measurement | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kyuhan Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (3):
- South Korea (3):
  - Chung-ang University Hospital, Seoul
  - Konkuk University Hospital, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No